CLINICAL TRIAL: NCT01788735
Title: Unexplained Infertility Among Asthmatic and Atopic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Elisabeth Juul Gade (Other)
Collaborators: Danish Medical Association (Other)
Responsible Party: Sponsor-Investigator, Elisabeth Juul Gade, MD, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Other Study IDs: AF
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Atopics; Unexplained Infertility
Keywords: unexplained infertility; asthma; allergy
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blod, serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Unexplained infertility is defined as the lack of thec ability to become pregnant during the first year, although the periods of the woman, the semen from the man and the laparoscopic findings are normal. In Denmark do roughly every fifth to seven couple in the fertile age have problems becoming pregnant for a various kind of reasons, of these are 10-15 % unexplained infertile.

Many factors are pointed out as imported. In particularly lifestyle factors such as the diet, smocking, obesity, lack of physic activity and alcohol. The causal connection is yet to be found, but it is assumed that there is a link between infertility and endocrine, neurological and immunological factors.

Asthma and allergy are some of the most common diseases among young people in western world .The development of these diseases are caused by both hereditary factors, and factors that also seem to be important in infertility.

It is clinically observed that many unexplained infertile patients simultaneously suffer from asthma and allergy. Furthermore this group of patients seems harder to treat in terms of becoming pregnant during fertility treatment then healthy not asthmatic and non allergic persons.

There is limited available data about this subject and the data that is already collected does not show a clear tendency.

Hypothesis: Atopic asthma is characterized by a systemic inflammation and can therefore be the reason for infertility among this group of patients.

The aim:

The aim of this study is to examine whether female asthmatics and allergic are less fertile then healthy females- whether there is there a link between asthma and infertility. Furthermore if an optimal asthma treatment during fertility treatment reduces time to pregnancy.

DETAILED DESCRIPTION:
Introduction:

Unexplained infertility is defined as the lack of thec ability to become pregnant during the first year, although the periods of the woman, the semen from the man and the laparoscopic findings are normal. In Denmark do roughly every fifth to seven couple in the fertile age have problems becoming pregnant for a various kind of reasons, of these are 10-15 % unexplained infertile.

Many factors are pointed out as imported. In particularly lifestyle factors such as the diet, smocking, obesity, lack of physic activity and alcohol. The causal connection is yet to be found, but it is assumed that there is a link between infertility and endocrine, neurological and immunological factors.

Asthma and allergy are some of the most common diseases among young people in western world .The development of these diseases are caused by both hereditary factors, and factors that also seem to be important in infertility.

It is clinically observed that many unexplained infertile patients simultaneously suffer from asthma and allergy. Furthermore this group of patients seems harder to treat in terms of becoming pregnant during fertility treatment then healthy not asthmatic and non allergic persons.

There is limited available data about this subject and the data that is already collected does not show a clear tendency.

Hypothesis: Atopic asthma is characterized by a systemic inflammation and can therefore be the reason for infertility among this group of patients.

The aim:

The aim of this study is to examine whether female asthmatics and allergic are less fertile then healthy females- whether there is there a link between asthma and infertility. Furthermore if an optimal asthma treatment during fertility treatment reduces time to pregnancy.

The design:

The project is divided into 3 parts:

1. A Study of Population. In the first part of this project the aim is to evaluate the occurrence of asthmatic and allergic diseases among women with respectively normal fertility and infertility. This is done through data already collected in The Danish twin Study from 1998- 2002 concerning questions about asthma, hay fever, atopic eczema and number of children.
2. A Prospective Study In the second part of this project the aim is to examine clinically, whether female asthmatics in general have more difficulties becoming pregnant then non- asthmatic females. Furthermore we aim to evaluate whether it is allergic or non allergic asthma that affects the fertility the most.
3. Casual study In the third part of this project we only include 40 of the unexplained infertile females collected earlier- 10 females with asthma, 10 females with allergy, 10 females with both asthma and allergy, 10 without any atopic disease.These women have, in addition to the initial asthma and allergy diagnosis, made a suction of the mucus in the uterus, when they are ovulating. This in order to determine whether the environment in the uterus is different in terms of inflammation in atopics. The aim of this study is to find an explanation for a possible decreased pregnancy rate and a longer time to pregnancy in atopics.

Material :

396 unexplained infertile females are included, when starting treatment at a fertility clinic. Among these are 197 healthy unexplained infertile females and 197 are females with the combination asthma and unexplained infertility. They are all included due to specific inclusion and exclusion criteria.

Methods:

All subjects are by inclusion tested for asthma with bronchial provocation tests. The pulmonary function is measured and the severity of their possible asthma is examined by NO in the expired air. Blood samples (RAS test) and prick test are performed to evaluate their possible allergy status. All subjects are to fill out questionnaires concerning asthma, allergy and their infertility. Due to the test mentioned above the subjects are divided in to groups, asthmatic , allergics, atopics and non- atopics.

The female asthmatics are treated due to the international guidelines. All groups are followed till achieved pregnancy; where after time to pregnancy can be compared.¨

In the third part of the study a suction of the mucus in the uterus is made at time of ovulation, to determinate the level of inflammation in atopics versus non atopics at time of fertilization.The mucus is examined fore inflammatory markers related to atopy such as TNF alpha, IL4,5,6,8and 33.

ELIGIBILITY:
Inclusion Criteria:

* unexplained infertile

Exclusion Criteria:

* no other diseases of the lung then asthma
* non- smoking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young healthy wemon that are unexplained infetile and have asthma, atopic ezcema or allergy
Sampling Method: Probability Sample
Enrollment: 396 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Time to pregnancy | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, Professor, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Respiratory Research Unit, Bispebjer Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Gade EJ, Thomsen SF, Lindenberg S, Backer V. Fertility outcomes in asthma: a clinical study of 245 women with unexplained infertility. Eur Respir J. 2016 Apr;47(4):1144-51. doi: 10.1183/13993003.01389-2015. Epub 2016 Feb 11. PMID 26869675